CLINICAL TRIAL: NCT00131638
Title: Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Weekly Doses of Palifermin (rHuKGF) for the Reduction of Oral Mucositis in Subjects With Advanced Head and Neck Cancer Receiving Adjuvant Radiotherapy and Chemotherapy(RT/CT)
Brief Title: A Study of Palifermin for the Reduction of Oral Mucositis in Subjects With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20040118
Record Dates: First submitted 2005-07-26; First posted 2005-08-19 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: Oncology; KGF; Palifermin; Oral mucositis; Clinical Trial; Amgen; head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Stomatitis | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palifermin (Experimental): Single IV dose of palifermin at 120 μg/kg, 3 days before the start of radiotherapy plus 6 once weekly palifermin doses at the same dose level during a 6-week Radiotherapy / chemotherapy course
  Interventions: Drug: Palifermin
- Placebo (Placebo Comparator): Single IV dose of placebo at 120 μg/kg, 3 days before the start of Radiotherapy, plus 6 once weekly placebo doses at the same dose during a 6-week radiotherapy / chemotherapy course.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Single IV dose of placebo at 120 μg/kg, 3 days before the start of Radiotherapy, plus 6 once weekly placebo doses at the same dose during a 6-week radiotherapy / chemotherapy course.
  Other Names: Pbo
  Arms: Placebo
Drug: Palifermin — Single IV dose of palifermin at 120 μg/kg, 3 days before the start of radiotherapy plus 6 once weekly palifermin doses at the same dose level during a 6-week Radiotherapy / chemotherapy course
  Other Names: KGF
  Arms: Palifermin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of palifermin (recombinant human keratinocyte growth factor, rHuKGF) in reducing the incidence of severe oral mucositis in subjects with locally advanced head and neck cancer receiving radiotherapy with concurrent chemotherapy as adjuvant treatment for their disease.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the efficacy of palifermin administered intravenously (IV) in weekly doses (minimum of 7 weekly doses, until RT was complete) in reducing the incidence of severe (World Health Organization [WHO] grade 3 or 4) oral mucositis in subjects with locally advanced HNC receiving RT concurrent with CT (RT/CT) as adjuvant treatment for their disease (postoperative setting). This study will assess the safety and tolerability of palifermin at the dose of 120 μg/kg IV administered weekly (minimum 7 weekly doses, until RT was complete) in this subject population. This study will also evaluate the effect of palifermin on the clinical sequelae of severe OM (eg, average subject-reported mouth and throat soreness [MTS] score), and on RT-induced xerostomia in this population, as well as the long-term effects of palifermin on disease outcome and survival in this population.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented squamous cell carcinoma ( AJCC [American Joint Committee on Cancer] Stage II, III, IVA or IVB) involving either the oral cavity, oropharynx, hypopharynx, or larynx,post surgical resection (R0, R1) and candidates for adjuvant RT/CT
* Radiation treatment field to receive planned dose of at least 50Gy to area of the oral cavity/oropharynx mucosa that can be visualized
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Functional hematopoietic and hepato-renal systems

Exclusion Criteria:

* Tumors of the lips, paranasal sinuses, salivary glands, or unknown primary tumors
* Metastatic disease (M1) Stage IV C
* Presence or history of any other primary malignancy (other than curatively treated in situ cervical cancer or basal cell carcinoma of the skin)
* History of chronic pancreatitis or episode of acute pancreatitis within the last year
* Prior radiation to the site of the disease, or prior chemotherapy-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence percentage of severe oral mucositis (Grades 3 or 4 on the WHO oral mucositis scale) | Up to 24 weeks

SECONDARY OUTCOMES:
Average patient-reported mouth and throat soreness score (as reported on Question 3 of the Oral Mucositis Weekly Questionnaire for patients with Head and Neck cancer [OMWQ-HN] | 16 weeks
Time to onset of severe oral mucositis (WHO Grades 3 or 4) | 12 weeks
Total dose of opioid analgesics used (mg of morphine equivalents) | 16 weeks
Incidence of unplanned delays in CT for cisplatin administration on Day 22 (to include discontinuations of CT) | 12 weeks
Incidence of xerostomia (CTCAE v3.0 Dry Mouth/Xerostomia scale Grade 2 or higher) | 10 years
Duration of severe oral mucositis (WHO Grades 3 or 4) | 15 weeks
Incidence of >/equal to 5 missed consecutive fractions of scheduled RT (to include discontinuations of RT) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Henke M, Alfonsi M, Foa P, Giralt J, Bardet E, Cerezo L, Salzwimmer M, Lizambri R, Emmerson L, Chen MG, Berger D. Palifermin decreases severe oral mucositis of patients undergoing postoperative radiochemotherapy for head and neck cancer: a randomized, placebo-controlled trial. J Clin Oncol. 2011 Jul 10;29(20):2815-20. doi: 10.1200/JCO.2010.32.4103. Epub 2011 Jun 13. PMID 21670447
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_24_KGF_20040118.pdf
- See also: FDA-approved Drug Labeling — http://www.kepivance.com/